CLINICAL TRIAL: NCT00521911
Title: Detection and Treatment of Depression in Patients Admitted to the General Hospital
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Radboud University Medical Center (Other)
Responsible Party: Anne EM Speckens, PhD, MD, Radboud University Medical Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PROJECT9999
Record Dates: First submitted 2007-08-27; First posted 2007-08-28 (Estimated); Last update posted 2008-12-25 (Estimated); Status verified 2008-12

CONDITIONS: Depressive Disorder; Depression
Keywords: Intervention Studies; Randomized Controlled Trials; Cognitive Therapy; Hospitals, General; Prevalence
MeSH Terms: conditions — Depressive Disorder; Depression | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator): Cognitive Behavioural Therapy
  Interventions: Behavioral: Cognitive Behavioural Therapy
- 2 (No Intervention): Treatment as Usual

INTERVENTIONS:
Behavioral: Cognitive Behavioural Therapy
  Arms: 1

SUMMARY:
Depression is a common disorder among patients with a somatic illness admitted to the general hospital. Patients with depression do worse in terms of their somatic symptoms or functioning that those without depression. They also stay in the hospital for longer.

That is the reason that we are interested to know whether patients with depression do better if their depression is recognised earlier and treated appropriately. We would like to find out which questionnaires are most suitable in clinical practice to help pick up patients with a depression. In addition, we would like to know whether a short-term psychological treatment of depression would be of any help. We hope to be able to show that this treatment would not only result in a reduction of depressive symptoms, but also in a better and quicker recovery of the somatic illness.

The treatment will consist of 6 to 9 weekly sessions of one hour, conducted by a cognitive behavioural assistant. Initially, the treatment will take place in the hospital. When patients are discharged, treatment sessions will continue at home. The treatment will focus on things like recognising and challenging unhelpful thoughts, planning of activities, and testing out of predictions by setting up behavioural experiments. Three monthly booster sessions will be offered to help patients to maintain their gains and prevent relapse. We will reassess the symptoms of the patients at three and six months after the end of treatment.

ELIGIBILITY:
Inclusion Criteria:

* Depressive Disorder

Exclusion Criteria:

* Severe Physical Disfunction
* Severe Cognitive Disfunction
* Speech and/or Hearing Disorder
* Limited knowledge of the Dutch language

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2007-08; Primary Completion 2008-12 (Estimated); Study Completion 2008-12 (Estimated)

PRIMARY OUTCOMES:
Depressive Disorder Physical symptoms | 9 months

SECONDARY OUTCOMES:
- Functional impairment (RAND 36) - Cost-effectiveness (TiC-P) - Quality of Life (EQ5D) | 9 months

CONTACTS AND LOCATIONS:
Overall Officials: Anne EM Speckens, PhD, MD, Principal Investigator — Radboud University Medical Center
Locations (1):
- Radboud University Nijmegen Medical Centre, Nijmegen, Gelderland, Netherlands

REFERENCES:
- See also: Radboud University Nijmegen Medical Centre — http://www.umcn.nl